## Feasibility and Preliminary Effects of using a Music-based, Rhythm-modulating Wearable Sensor System in the Community in Persons With Parkinson Disease

Statistical Analysis Plan

NCT Number: NCT04891107

Date of Document: July 27, 2023

## TEMPO Statistical Analysis Plan

Normality of distribution will be confirmed using Shapiro-Wilk test. Given the preliminary nature of this study, adjustments are not planned to account for multiple comparisons across outcomes.

## **Primary Outcomes:**

- >Feasibility metrics will be measured descriptively
- >PDQ-39 mobility dimension will be assessed using paired t-tests ( $\alpha$  = .05) to compare baseline and post-intervention values

## Secondary Outcomes:

- > Change in disease severity (MDS-UPDRS III), walking endurance (6MWT), gait speed (10MWT), change in mobility (FTSTS) and overall quality of life (PDQ-39 total score) will be assessed using paired t-tests ( $\alpha$  = .05) to compare baseline and post-intervention values.
- >Change in daily steps and moderate intensity minutes will be assessed using paired t-tests ( $\alpha$  = .05) to compare daily walking activity at baseline (days 1-4) to daily walking activity during the intervention (days 5-8).